CLINICAL TRIAL: NCT04637074
Title: Registrated Cohort Study on Thrombectomy for Stroke
Brief Title: A Cohort Study on Thrombectomy for Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ning Wang, MD., PhD. (Other)
Responsible Party: Sponsor-Investigator, Ning Wang, MD., PhD., Director of Neurology department, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA, ECFAH of FMU [2020]389
Record Dates: First submitted 2020-11-15; First posted 2020-11-19 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10mL venous blood sample will be collected Each participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The cerebral collateral circulation refers to the subsidiary network of vascular channels that stabilize cerebral blood flow when principal conduits fail. Collateral status differs among patients with acute ischemic stroke. Relatively sparse attention has been devoted to the role of baseline collateral circulation in patients with acute ischemic stroke who are candidates for revascularization. This study aim to investigate the correlation between baseline collateral circulation and the likelihood of opening of an arterial occlusion, the extent of reperfusion, tissue injury and clinical impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Mechanical thrombectomy initiated within 24 hours after onset
* CT perfusion can be performed before the initiation of thrombectomy and 24h after thrombectomy

Exclusion Criteria:

* Contraindication to imaging with contrast agents
* Delay between imaging and beginning of thrombectomy > 90 minutes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients experiencing brain infarction complicating the large-vessel occlusion
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale | 3 month
  Good functional outcome will be defined by a Modified Rankin Scale of 0-2, 3 months after stroke onset

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, First Affiliated Hospital of Fujian Medical University, Fuzhou, China